CLINICAL TRIAL: NCT04872439
Title: Novel Antineuronal Antibodies in Gastrointestinal Motility Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00114555
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Gastrointestinal Dysmotility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum isolated from blood, DNA isolated from blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Antibody isolation, DNA isolation: Patients with GI dysmotility
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Patients with autoimmune gastrointestinal dysmotility will provide 20 mL of blood to isolate serum, plasma and peripheral blood mononuclear cells for whole exome sequence. Antibodies to be isolated are: Antineuronal nuclear antibody type 1,Collapsing response-mediator family immunoglobulin G, Ganglionic Acetylcholine Receptor Antibody, Muscle Acetylcholine Receptor Antibody, Striational, Voltage-gated calcium channel, N- type, Voltage-gated calcium channel, P/Q- type, Voltage-gated potassium channel, Glutamic Acid Decarboxylase 65, Gastric parietal cell, Thyroperoxidase, Thyroglobulin

SUMMARY:
Gastrointestinal motility disorders represent a heterogeneous group of neuromuscular diseases of the enteric nervous systems. While autoimmune neuromuscular diseases of the central nervous system (CNS) are well described, the role of autoimmunity in enteric nervous system (ENS) has been less studied. Approximately 10% of patients with unexplained gastrointestinal dysmotility diseases have positive serum autoantibodies to peripheral nervous system proteins, suggesting an autoimmune mechanism targeting the enteric nervous system. The investigator's aim is to identify novel anti neuronal antibodies that contribute to autoimmune gastrointestinal motility disorders by analyzing the serum of patients with abnormal gastrointestinal motility.

DETAILED DESCRIPTION:
Autoimmune gastrointestinal dysmotility (AGID) represents a subset of autoimmune disorders that affect the motor function of the gastrointestinal tract. It will often result in refractory gastrointestinal symptoms and poor quality of life. Approximately 10% of patients with unexplained gastrointestinal dysmotility diseases have positive serum autoantibodies to peripheral nervous system gangliosides and glycoproteins, which may be suggestive of an autoimmune mechanism targeting the enteric nervous system. The diagnosis is often made clinically in patients with gastrointestinal dysmotility in the context of primary autoimmune disease or a paraneoplastic syndrome. To date, specific diagnostic tests for AGID disorders do not exist. This study will aim to find whether patients with symptomatic autoimmune gastrointestinal dysmotility (AGID) will have a specific antigen and/or antibody causing the symptoms. The study will also aim to find whether patients with positive autoantibody titers will frequently have positive tilt-table testing (autonomic dysfunction).

The goal of this study is to determine the prevalence of autoimmune antibodies in patients presenting with unexplained GI dysmotility and refractory symptoms, and to examine the outcome (safety, tolerability, and clinical improvement) in a pilot cohort of such patients with a serum screening for antigens, antibodies, and validated questionnaires. This will be a prospective pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >13 years old.
* Patient referred to the GI Motility clinic for suspected enteric dysmotility based on chronic refractory gastrointestinal symptoms
* English proficiency and literacy sufficient to sign consent.

Exclusion Criteria:

* Pregnancy documented with a serum or urine pregnancy test. If participants believe that they are pregnant, they will need to notify a study physician who will order a serum or urine test for pregnancy and remove them from the study if the test results come back positive.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with autoimmune gastrointestinal dysmotolity
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Antibodies for Autoimmune Gastrointestinal Dysmotility | Baseline
  Presence or absence of Autoimmune Gastrointestinal Dysmotility specific antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Ken J Hui, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States